CLINICAL TRIAL: NCT04720677
Title: Psychometric Properties of Adapted Turkish Version of ISYQOL Questionnaire in Patients With AIS
Status: Completed | Type: Observational
Sponsor: Hürriyet Yılmaz (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor-Investigator, Hürriyet Yılmaz, MD.Prof., Halic University
Organization: Halic University (Other)
Other Study IDs: HUEK172-31
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Adolescent Idiopathic Scoliosis; Health Related Quality of Life
Keywords: Adolescent Idiopathic Scoliosis; Quality of Life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish Version of The Italian Spine Youth Quality of Life (ISYQOL) Questionnaire — Turkish Version of The Italian Spine Youth Quality of Life (ISYQOL) Questionnaire

SUMMARY:
The ISYQOL questionnaire was translated into Turkish and was assessed the psychometric properties of the Turkish version of the ISYQOL in terms of test-retest reliability, internal consistency, and construct validity in this research.

DETAILED DESCRIPTION:
HRQOL is considered one of the most relevant outcomes of both conservative and surgical treatment of scoliosis, for this reason, several questionnaires (e.g. SRS-24 and SRS-22) have been developed. SRS-22 has been reported as the most commonly used scale to measure HRQOL in patient with scoliosis in many countries. However, current literature showed that SRS-22 has poor measurement properties, it does not satisfy fundamental measure requirements, i.e. additivity, generalizability and unidimensionality. According to Rasch analysis study SRS-24 and SRS-22 presents high ceiling effects in conservative care, for the reason that was developed for surgical candidates. The Italian Spine Youth Quality of Life (ISYQOL) questionnaire originally in Italian, is the first HRQOL questionnaire developed according to the Rasch analysis. It was developed in a conservative treatment setting for all type of spinal deformities, including also patients with surgical curves. The ISYQOL has recently been translated into English, however, its adaptation to the Turkish language is necessary for use in the Turkish population. The psychometric properties of any scale may be affected by translation into another language, that's why it is important for the scale to be evaluated psychometrically. Therefore, the purpose of this study was to translate the ISYQOL questionnaire to Turkish and to assess the psychometric properties of the Turkish version of the ISYQOL in terms of test-retest reliability, internal consistency and construct validity when used on patients with idiopathic scoliosis. Adolescent girls with idiopathic scoliosis who applied to Formed Scoliosis Treatment and Brace Center between September 2018 to 2020 are inviting in this stud by mailing

ELIGIBILITY:
Inclusion Criteria:

* who has diagnosed with AIS
* aged 10 to 18 years
* curvature between 10 ° to 45 ° ,
* native Turkish speaker adolescents who accepted to participate in the study and approved by their parents.

Exclusion Criteria:

* non-idiopathic scoliosis
* history of spinal surgery,
* spinal trauma, tumor, infection

Ages: 10 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Investigators could not analyze the sex-related difference in this study. In clinical practice, investigators have more female cases and they could not reach a male sample large enough to compare with them.
Study Population: Adolescent girls with idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Turkish Version of The Italian Spine Youth Quality of Life (ISYQOL) Questionnaire | baseline
  ISYQOL, is a 20-item tool used to assess spine health and health related quality of life in patients with spinal deformities. ISYQOL was developed according to Rasch analysis. Seven ISYQOL items assess the impact of bracing on quality of life and are to be administered only to people wearing the brace. Because of ISYOQL is a Rasch-consistent questionnaire, it allows the comparison of the HRQOL in AIS patients who wearing and not wearing the brace. Each item is rated on a 0-2 point Likert scale from never to often. Total scores range from 0 to 40. Lower scores on the ISYQOL indicate higher health-related quality of life
SRS-22 Patient Questionnaire | baseline
  SRS-22 questionnaire was developed by SRS to evaluate health-related quality of life (HRQL) in patients with adolescent idiopathic scoliosis (AIS) and the Turkish version was validated in 2005. The SRS-22 questionnaire consists of 22 items Likert type scale that allows scoring between 1-5 for each question. SRS-22 has five domains including function, pain, mental health, self-image and satisfaction. Subgroups can be evaluated separately, or the total score is obtained by summing up the scores from all questions. The total score of each section ranges from 5 to 25, only the section evaluating satisfaction from the treatment is in the range of 2-10. Scoring is obtained by dividing the total score of each section by the number of questions in that section. Higher scores indicate better quality of life.
Re-Test Reliability of Turkish Version of ISYQOL Questionnaire | 4 weeks after from the first assessment
  Test-retest reliability was assessed by calculating the intraclass correlation coefficient (ICC).ICC interpreted; proposed a classification for the strength of test-retest reliability based on the ICC as follows: less than 0.40 is poor, between 0.40-0.75 is fair to good and; more than 0.75 is excellent.

SECONDARY OUTCOMES:
Cobb angle | baseline
  Cobb angle is determinant of curvature severity which obtain from full spine PA radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen Büyükaslan, PT,PhD(c), Principal Investigator — Medipol University; Hürriyet Yılmaz, MD, Prof., Study Director — Halic University; Melek Güneş Yavuzer, MD, Prof., Study Director — Halic University
Locations (1):
- Formed Healthcare Scoliosis Brace and Treatment Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No